CLINICAL TRIAL: NCT01817751
Title: Phase 2 Study of Sorafenib, Valproic Acid, and Sildenafil in the Treatment of Recurrent High-Grade Glioma
Brief Title: Sorafenib, Valproic Acid, and Sildenafil in Treating Patients With Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14816; HM14816 (Other: VCU IRB); NCI-2013-00705 (Other: NCI); P30CA016059 (NIH)
Record Dates: First submitted 2013-03-20; First posted 2013-03-25 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Glioblastoma; Recurrent Adult Brain Neoplasm; Malignant Glioma; WHO Grade III Glioma
Keywords: central nervous system; Brain and Nervous System
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma; Neurologic Manifestations | interventions — Sorafenib; Valproic Acid; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (sorafenib tosylate, valproic acid, sildenafil) (Experimental): * Sorafenib 400 mg orally twice a day;
  * Valproic acid (to levels ≥ Lower Level of Normal (LLN) orally twice a day;
  * Sildenafil 50 mg orally twice a day
  A cycle consists of 4 weeks.
  *The first 6 patients evaluable for qualifying toxicity assessment will be treated as a safety lead-in; enrollment will be gated (the first 3 evaluable patients must complete 4 weeks of the combination therapy before the next 3 patients start combination treatment on protocol)
  Interventions: Drug: sorafenib tosylate; Drug: valproic acid; Drug: sildenafil citrate

INTERVENTIONS:
Drug: sorafenib tosylate — Given by mouth
  Other Names: pyridinecarboxamide, chloro-trifluoromethylphenyl pyridine-carboxylic acid methylamide-methylbenzenesulfonate tosylate, Nexavar
Drug: valproic acid — Given by mouth
  Other Names: 2-Propylpentanoic or Propylvaleric Acid, Alti-Valproic, Depakene, Di-n-propylacetic Acid, Ergenyl, Novo-Valproic, VA, Valproate, Valproate Sodium
Drug: sildenafil citrate — Given by mouth
  Other Names: Viagra

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of the combination of three drugs, sorafenib (Nexavar®), valproic acid (Depakote®), and sildenafil (Viagra®), when used to treat high-grade glioma, a type of brain tumor.

DETAILED DESCRIPTION:
The study is a single-center, open-label phase 2 study, with an early stopping rule in place for safety. The trial will include patients with recurrent or progressive high-grade glioma.

The trial will be conducted in an adaptive design, with a Simon's mini-max 2-stage design incorporating an interim analysis for efficacy

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed high-grade glioma (World Health Organization (WHO) grade 3 or 4), with documented computed tomography (CT) or magnetic resonance imaging (MRI) progression or recurrence. Biopsy is also an acceptable method of confirming progression or recurrence. If initial tumor was grade 2 glioma, histological confirmation of high-grade recurrence is required

  * After first interim analysis, if the study proceeds to enrollment of selected patients (only those who have platelet-derived growth factor receptor (PDGFRa)-positive tumors), patients will be pre-registered for PDGFRa analysis and registered to the combination treatment schema only if PDGFRa-positive an all other enrollment criteria are met.
* Measurable or evaluable disease by response assessment in neuro-oncology (RANO) (MRI) or MacDonald (CT) criteria
* Fixed or decreasing dose of corticosteroids (or no corticosteroids) for at least 1 week prior to cycle 1 day 1.
* At least 12 weeks since the completion of radiation therapy to a total of >=50 Gray (Gy).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* White blood cell (WBC) >= 3,000/mm^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin (Hgb) >= 8.5 g/dL
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN) for the laboratory
* Total bilirubin =< 1.5 x ULN for the laboratory (total bilirubin criteria may be waived if a patient has documented Gilbert's disease)
* Creatinine clearance (CrCL) >= 30 mL/min as calculated by standard Cockcroft-Gault equation
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use a medically accepted form of birth control for the duration of study participation and for 2 months following completion of study treatment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Investigational agent within 4 weeks of first dose of study treatment
* Prior bevacizumab or tyrosine-kinase inhibitor
* History of allergic reactions or intolerance to any of the required agents on the study
* Any condition that would prohibit patient from initiating valproic acid. Current or prior valproic acid treatment is allowed (do not need to be ≥ LLN for laboratory for enrollment).
* Seizure disorder necessitating the use of enzyme-inducing antiepileptic drugs (EIAEDs). Efforts may be made by the treating physician to change the antiepileptic drug from another agent to valproic acid or non-EIAED prior to excluding the patient from study
* Contraindication to antiangiogenic agents, including:

  * Bronchopulmonary hemorrhage/bleeding event >= grade 2 (NCI Common Terminology Criteria for Adverse Events [CTCAE] version 4.0) within 4 weeks or less prior to first dose of study drug
  * Any other hemorrhage/bleeding event >= grade 3 (NCI CTCAE v4.0) within 4 weeks or less prior to first dose of study treatment
  * Radiological evidence of any intracranial hemorrhage within the 4 weeks or less less prior to first dose of study treatment
  * History of significant intratumoral, intracerebral, or subarachnoid hemorrhage
  * Serious non-healing wound, ulcer, or bone fracture
  * Documented bowel perforation within 6 months of the start of study treatment.
* Major surgery within 2 weeks of the start of study treatment, or ongoing complications from surgeries performed previously
* Clinically significant cardiac disease, including major cardiac dysfunction, such as uncontrolled angina, clinical congestive heart failure with New York Heart Association (NYHA) class III or higher, ventricular arrhythmias requiring antiarrhythmic therapy, recent (within 6 months) myocardial infarction or unstable coronary artery disease.
* Systolic blood pressure (BP) > 160 mm Hg or diastolic pressure > 100 mm Hg despite optimal medical management
* History of priapism
* Known history of retinitis pigmentosa
* Known mitochondrial disorder caused by mutations in mitochondrial DNA polymerase γ.
* Arterial thromboembolic or embolic events such as myocardial infarction, cerebrovascular accident, including transient ischemic attacks 6 months prior to first study treatment
* Serious uncontrolled infection > grade 2 (CTCAE v 4)
* Known human immunodeficiency virus (HIV) positivity
* Unable to swallow medication or suspected malabsorption
* Patients on chronic nitrate therapy or alpha-blockers

  * Exclude persons who require ongoing administration of STRONG CYP3A4 inhibitors and/or STRONG CYP3A4 inducers and/or STRONG CYP2C9 inhibitors.
* Women who are pregnant or nursing
* Persistent heart rate (HR) <50 or >120 beats per minute (bpm)
* Corrected QT (QTc) > 480 ms (grade 2 or greater) on screening electrocardiogram (ECG)

  * If baseline QTc on screening ECG meets exclusion criteria on screening assessment:
  * Check potassium and magnesium levels
  * Correct any identified hypokalemia and/or hypomagnesemia and repeat ECG to confirm exclusion of patient due to QTc
  * For patients with a heart rate (HR) 60-100 bpm, no manual read of QT is required
  * For patients with baseline HR < 60 or > 100 bpm, manual read of QT by cardiologist is required using Fridericia correction
* Other condition(s) that in the opinion of the investigator might compromise the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-04-11 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang F, Liu Y, Chou FJ, Yang C. Genotoxic therapy and resistance mechanism in gliomas. Pharmacol Ther. 2021 Dec;228:107922. doi: 10.1016/j.pharmthera.2021.107922. Epub 2021 Jun 23. PMID 34171339

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil): * Sorafenib 400 mg orally twice a day;
  * Valproic acid (to levels ≥ Lower Level of Normal (LLN) orally twice a day;
  * Sildenafil 50 mg orally twice a day
  A cycle consists of 4 weeks.
  *The first 6 patients evaluable for qualifying toxicity assessment will be treated as a safety lead-in; enrollment will be gated (the first 3 evaluable patients must complete 4 weeks of the combination therapy before the next 3 patients start combination treatment on protocol)
  sorafenib tosylate: Given by mouth
  valproic acid: Given by mouth
  sildenafil citrate: Given by mouth
Period: Overall Study
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Started | 47
Completed | 46
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 6-Month Progression Free Survival (PFS)
Description: Number of patients evaluable for response, regardless of tumor platelet derived growth factor receptor (PDGFR) status, with 6- month PFS defined as the time from the first day a patient receives study treatment until time of progression per response assessment in neuro-oncology (RANO) or Macdonald criteria or death, whichever occurs first.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 47
Participants
  Met 6 month PFS | 8
  Did not meet 6 month PFS | 25
  Not Evaluable | 14

2. Secondary Outcome: Number of Participants Whose Tumors Express PDGFRa With and Without 6-Month PFS.
Description: Number of patients evaluable for response, with tumors that express PDGFRα, with 6-month PFS defined as the time from the first day a patient receives study treatment until time of progression per RANO or Macdonald criteria or death, whichever occurs first.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 33
Participants
  Express PDGFRa that met 6 month PFS | 5
  Express PDGFRa that did not meet 6 month PFS | 7
  Did not express PDGFRa that met 6 month PFS | 2
  Did not express PDGFRa that did not met 6 months | 7
  Not evaluable | 12

3. Secondary Outcome: Number of Participants With Best Response of CR Plus Number of Participants With Best Response of PR.
Description: Overall response rate (CR+PR), using RANO or Macdonald criteria, in patients evaluable for response regardless of tumor PDGFR status
Time Frame: From the first day of study treatment until best response or off study, up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 47
Participants
  # Pts with best response of CR | 0
  # Pts with best response of PR | 1
  # Pts without best response of PR or CR | 32
  # Pts not evaluable | 14

4. Secondary Outcome: Number of Participants Whose Tumors Express PDGFRa With Best Response of CR Plus Number of Participants Whose Tumor Expresses PDGFRa With Best Response of PR.
Description: Overall response rate (CR+PR), using RANO or Macdonald criteria, in patients who are evaluable for response and who have tumors that express PDGFRα.
Time Frame: From initiation of study treatment to time of best response or off-study (up to 4 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 17
Participants
  # Pts with best response of CR | 0
  # Pts with best response of PR | 0
  # Pts without best response of PR or CR | 12
  # Pts not evaluable | 5

5. Secondary Outcome: Number of Participants With 12-Month Overall Survival (OS)
Description: Number of patients evaluable for response, regardless of tumor PDGFR status, who are alive at 12 months after the first day a patient receives study treatment. Overall Survival (OS) defined as the time from the first day a patient receives study treatment until death by any cause.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 47
Participants | 14

6. Secondary Outcome: Number of Participants Whose Tumors Express PDGFRa With and Without 12-Month OS.
Description: Number of patients evaluable for response with tumors that express PDGFRα who are alive at 12 months after the first day a patient receives study treatment. On study is defined as the time from the first day a patient receives study treatment until death by any cause.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 33
Participants
  Expressed PDGFRa with12 month OS | 6
  Expressed PDGFRa with less than 12 month survival | 6
  Negative for PDGFRa with 12 month OS | 3
  Negative for PDGFRa without 12 month OS | 6
  Not Evaluable | 12

7. Secondary Outcome: Evaluation of Safety and Toxicity of Sorafenib, Valproic Acid, and Sildenafil
Description: Number of patients with adverse events
Time Frame: From initiation of study therapy to completion of adverse event (AE) observation period, up to 30 days following the end of study treatment, up to 7 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
Number analyzed (Participants) | 47
Participants | 47

ADVERSE EVENTS:
Time Frame: From initiation of study therapy to completion of adverse event (AE) observation period, up to 30 days following the end of study treatment up to 7 years.
Description: Number of patients with adverse events, and types of events, as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI CTCAE v4.0).
Arm/Group | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil)
All-Cause Mortality (participants affected / at risk) | 1/47
Serious Adverse Events (participants affected / at risk) | 17/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil) (N=47)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
abdominal Pain (Gastrointestinal disorders) | 1 (1)
Colonic Perforation (Gastrointestinal disorders) | 1 (1)
ileal fistula (Gastrointestinal disorders) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 1 (1)
edema Limbs (Hepatobiliary disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
gait disturbance (General disorders) | 3 (3)
general disorders and administration site conditions (General disorders) | 1 (1)
multi-organ failure (General disorders) | 1 (1)
appendicitis (Infections and infestations) | 1 (47)
fall (Injury, poisoning and procedural complications) | 2 (2)
fracture (Injury, poisoning and procedural complications) | 1 (47)
alanine aminotransferase increased (Investigations) | 2 (2)
aspartate aminotransferase increased (Investigations) | 1 (1)
investigations-other, specify (Investigations) | 2 (2)
lipase increased (Investigations) | 1 (1)
neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (3)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
muscle weakness, right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
concentration impairment (Nervous system disorders) | 1 (1)
dysphasia (Nervous system disorders) | 2 (2)
hypersomnia (Nervous system disorders) | 1 (1)
lethargy (Nervous system disorders) | 1 (1)
seizure (Nervous system disorders) | 5 (6)
somnolence (Nervous system disorders) | 1 (1)
confusion (Psychiatric disorders) | 3 (3)
hematuria (Renal and urinary disorders) | 1 (1)
renal calculi (Renal and urinary disorders) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
social circumstances-other, specify (Social circumstances) | 1 (1)
hematoma (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate, Valproic Acid, Sildenafil) (N=47)
anemia (Blood and lymphatic system disorders) | 19 (22)
atrial fibrillation (Cardiac disorders) | 1 (1)
cardiac disorders-other, specify (Cardiac disorders) | 1 (1)
sinus bradycardia (Cardiac disorders) | 7 (8)
sinus tachycardia (Cardiac disorders) | 5 (5)
ear and labyrinth disorders-other, specify (Ear and labyrinth disorders) | 2 (2)
hearing impaired (Ear and labyrinth disorders) | 3 (3)
tinnitus (Ear and labyrinth disorders) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1)
cushingoid (Endocrine disorders) | 1 (1)
endocrine disorders-other, specify (Endocrine disorders) | 1 (1)
hyperthyroidism (Endocrine disorders) | 1 (1)
blurred vision (Eye disorders) | 8 (10)
eye disorders-other, specify (Eye disorders) | 5 (6)
eye pain (Eye disorders) | 1 (1)
watering eyes (Eye disorders) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 8 (12)
bloating (Gastrointestinal disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 7 (8)
diarrhea (Gastrointestinal disorders) | 21 (34)
dry mouth (Gastrointestinal disorders) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 4 (4)
dysphagia (Gastrointestinal disorders) | 4 (4)
fecal incontinence (Gastrointestinal disorders) | 7 (10)
flatulence (Gastrointestinal disorders) | 3 (3)
gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (9)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6 (7)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
mucositis oral (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 11 (12)
oral dysesthesia (Gastrointestinal disorders) | 2 (2)
oral hemorrhage (Gastrointestinal disorders) | 1 (1)
toothache (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 7 (8)
edema face (General disorders) | 1 (1)
edema limbs (General disorders) | 6 (9)
fatigue (General disorders) | 26 (34)
fever (General disorders) | 1 (1)
gait disturbance (Gastrointestinal disorders) | 13 (14)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3)
Generalized edema (General disorders) | 1 (4)
irritability (General disorders) | 1 (1)
malaise (General disorders) | 4 (4)
non-cardiac chest pain (General disorders) | 1 (1)
pain (General disorders) | 6 (12)
allergic reaction (Immune system disorders) | 2 (3)
eye infection (Infections and infestations) | 1 (1)
infections and infestations-other, specify (Infections and infestations) | 3 (3)
mucosal infection (Infections and infestations) | 2 (2)
nail infection (Infections and infestations) | 1 (1)
otitis media (Infections and infestations) | 1 (1)
papulopustular rash (Infections and infestations) | 1 (1)
pharyngitis (Infections and infestations) | 1 (1)
prostate infection (Infections and infestations) | 1 (1)
skin infection (Infections and infestations) | 3 (5)
soft tissue infection (Infections and infestations) | 1 (3)
urinary tract infection (Infections and infestations) | 2 (2)
bruising (Injury, poisoning and procedural complications) | 11 (19)
wound complication (Injury, poisoning and procedural complications) | 1 (1)
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 17 (23)
alkaline phosphatase increased (Investigations) | 3 (4)
aspartate aminotransferase increased (Investigations) | 16 (22)
blood bilirubin increased (Investigations) | 4 (6)
cholesterol high (Investigations) | 3 (3)
creatinine increased (Investigations) | 3 (3)
GGT increased (Investigations) | 1 (1)
hemoglobin increased (Investigations) | 1 (1)
investigations - other, specify (Investigations) | 8 (17)
lymphocyte count decreased (Investigations) | 22 (36)
neutrophil count decreased (Investigations) | 20 (33)
platelet count decreased (Investigations) | 32 (48)
weight gain (Investigations) | 2 (4)
weight loss (Investigations) | 6 (13)
white blood cell decreased (Investigations) | 22 (36)
anorexia (Metabolism and nutrition disorders) | 13 (16)
dehydration (Metabolism and nutrition disorders) | 4 (4)
glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 4 (5)
hyperkalemia (Metabolism and nutrition disorders) | 10 (12)
hypermagnesemia (Metabolism and nutrition disorders) | 4 (4)
hypernatremia (Metabolism and nutrition disorders) | 3 (4)
hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
hypoalbuminemia (Metabolism and nutrition disorders) | 20 (26)
hypocalcemia (Metabolism and nutrition disorders) | 26 (41)
hypoglycemia (Metabolism and nutrition disorders) | 4 (7)
hypokalemia (Metabolism and nutrition disorders) | 13 (28)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (10)
hyponatremia (Metabolism and nutrition disorders) | 14 (19)
hypophosphatemia (Metabolism and nutrition disorders) | 35 (63)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
back pain (Musculoskeletal and connective tissue disorders) | 4 (7)
buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (13)
joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (2)
muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 (2)
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (4)
muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (3)
muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (8)
myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
cognitive disturbance (Nervous system disorders) | 3 (4)
concentration impairment (Nervous system disorders) | 3 (3)
depressed level of consciousness (Nervous system disorders) | 4 (4)
dizziness (Nervous system disorders) | 5 (6)
dysarthria (Nervous system disorders) | 2 (2)
dysesthesia (Nervous system disorders) | 1 (1)
dysgeusia (Nervous system disorders) | 7 (8)
dysphasia (Nervous system disorders) | 7 (8)
edema cerebral (Nervous system disorders) | 1 (1)
encephalopathy (Nervous system disorders) | 1 (1)
facial muscle weakness (Nervous system disorders) | 1 (1)
headache (Nervous system disorders) | 12 (19)
hypersomnia (Nervous system disorders) | 2 (2)
intracranial hemorrhage (Nervous system disorders) | 3 (3)
ischemia cerebrovascular (Nervous system disorders) | 1 (2)
lethargy (Nervous system disorders) | 7 (11)
memory impairment (Nervous system disorders) | 7 (8)
nervous system disorders- other, specify (Nervous system disorders) | 8 (9)
paresthesia (Nervous system disorders) | 4 (4)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
presyncope (Nervous system disorders) | 1 (1)
seizure (Nervous system disorders) | 5 (5)
sinus pain (Nervous system disorders) | 1 (1)
somnolence (Nervous system disorders) | 5 (6)
spasticity (Nervous system disorders) | 2 (2)
tremor (Nervous system disorders) | 4 (4)
Agitation (Psychiatric disorders) | 6 (7)
anxiety (Psychiatric disorders) | 5 (6)
confusion (Psychiatric disorders) | 15 (18)
delusions (Psychiatric disorders) | 1 (1)
depression (Psychiatric disorders) | 2 (3)
hallucinations (Psychiatric disorders) | 3 (4)
insomnia (Psychiatric disorders) | 8 (9)
personality change (Psychiatric disorders) | 1 (1)
psychiatric disorders- other, specify (Psychiatric disorders) | 1 (1)
suicidal ideation (Psychiatric disorders) | 1 (1)
hematuria (Renal and urinary disorders) | 5 (5)
proteinuria (Renal and urinary disorders) | 4 (5)
renal calculi (Renal and urinary disorders) | 1 (1)
urinary frequency (Renal and urinary disorders) | 6 (7)
urinary incontienence (Renal and urinary disorders) | 9 (11)
urinary retention (Renal and urinary disorders) | 2 (2)
urinary tract pain (Renal and urinary disorders) | 1 (1)
urinary urgency (Renal and urinary disorders) | 3 (3)
genital edema (Reproductive system and breast disorders) | 1 (1)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 5 (6)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (8)
alopecia (Skin and subcutaneous tissue disorders) | 7 (8)
body odor (Skin and subcutaneous tissue disorders) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 8 (9)
pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 20 (55)
pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
purpura (Skin and subcutaneous tissue disorders) | 2 (2)
rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 (22)
scalp pain (Skin and subcutaneous tissue disorders) | 4 (4)
skin and subcutaneous tissue disorders- other, specify (Skin and subcutaneous tissue disorders) | 10 (24)
skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
flushing (Vascular disorders) | 17 (18)
hematoma (Vascular disorders) | 1 (1)
hypertension (Vascular disorders) | 19 (44)
hypotension (Vascular disorders) | 3 (3)
thromboembolic event (Vascular disorders) | 2 (2)
fall (Injury, poisoning and procedural complications) | 12 (24)
fracture (Injury, poisoning and procedural complications) | 1 (3)
injury, poisoning and procedural complications- other, specify (Injury, poisoning and procedural complications) | 3 (3)
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT01817751/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT01817751/ICF_001.pdf